CLINICAL TRIAL: NCT07250841
Title: Cervical Intraepithelial Neoplasia Screening by Liquid-Based Pap Smear in General Gynecological Services Among Egyptian Women
Brief Title: Cervical Intraepithelial Neoplasia Screening Using Liquid-Based Pap Smear Among Egyptian Women
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tamer Abdelhamid Ahmed Abdelmaksoud, Obstetrics and Gynecology Resident, Kasr El Aini Hospital
Other Study IDs: MS-492025
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer (Early Detection)
Keywords: Liquid-Based Cytology; Pap Smear; Cervical Screening; HPV; CIN; Cervical Dysplasia; Bethesda System; Gynecological Screening; Egypt
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecological Screening: Women aged 25-60 attending Kasr Al-Aini outpatient gynecology clinics who undergo liquid-based Pap smear screening for detection of cervical intraepithelial neoplasia.
  Interventions: Diagnostic Test: Liquid-Based Pap Smear (LBC)

INTERVENTIONS:
Diagnostic Test: Liquid-Based Pap Smear (LBC) — Cervical sample collected using a cervical brush or broom and preserved in liquid fixative solution. Slides prepared using ThinPrep liquid-based cytology and reported according to the 2014 Bethesda System. Used for detection of abnormal cervical cytology including ASC-US, LSIL, HSIL, and NILM.

SUMMARY:
This observational study aims to screen Egyptian women aged 25-60 for cervical intraepithelial neoplasia (CIN) using liquid-based Pap smear during routine gynecological visits at Kasr Al-Aini outpatient clinics. Screening is performed through standardized liquid-based cytology to detect early cellular abnormalities that may indicate precancerous changes or cervical cancer. The goal of the study is to identify abnormal cytology at an early stage, improve early detection of cervical cancer, and provide epidemiological data on cervical abnormalities among women attending general gynecological services.

DETAILED DESCRIPTION:
This cross-sectional observational study was conducted at the Kasr Al-Aini outpatient gynecology clinics, Cairo University. A total of 984 women aged 25-60 years attending routine gynecologic care were enrolled after providing written informed consent. Women with pregnancy, prior hysterectomy, or known cervical lesions requiring diagnostic management were excluded.

Each participant completed a structured interview covering demographic characteristics, reproductive and sexual history, comorbidities, contraception use, and family history of malignancy. A standardized pelvic examination was performed, followed by cervical sampling using a cervical brush or broom. All samples were collected using the liquid-based cytology (LBC) technique, immediately preserved in fixative solution, and processed in the cytopathology laboratory using the ThinPrep system.

Slides were examined by experienced cytopathologists and classified according to the 2014 Bethesda System. Cytology results were categorized as NILM, ASC-US, LSIL, HSIL, or unsatisfactory. The primary objective was to detect any cytological abnormality suggestive of cervical intraepithelial neoplasia. Secondary objectives included describing the demographic and clinical correlates of abnormal cytology and estimating the overall prevalence of abnormal cervical cytology in this population.

The study aims to support earlier detection of cervical abnormalities, reduce progression to invasive cervical cancer, and provide population-based data to guide cervical cancer prevention strategies in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 25-60
* Attending Kasr Al-Aini outpatient gynecology clinics
* Willing to provide informed consent

Exclusion Criteria:

* • Pregnancy

  * Prior hysterectomy
  * Existing cervical lesions
  * Previous CIN treatment in last 5 years

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as female are eligible to participate, as the study involves cervical cytology screening and requires the presence of a cervix.
Study Population: Women aged 25-60 attending Kasr Al-Aini outpatient gynecology clinics and undergoing routine cervical screening using liquid-based cytology.
Sampling Method: Non-Probability Sample
Enrollment: 984 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Detection of Cervical Cytological Abnormalities | At time of screening (single visit)
  Presence of cytological abnormalities detected using liquid-based cytology (ThinPrep) and interpreted according to the 2014 Bethesda System.
  Unit of measure:
  Percentage of participants
  Outcome measure tool:
  Liquid-based cytology (LBC) using ThinPrep; Bethesda System classification (ASC-US, LSIL, HSIL, NILM, Unsatisfactory).

SECONDARY OUTCOMES:
Prevalence of Abnormal Cervical Cytology | At time of screening
  Proportion of screened women found to have abnormal cytology (ASC-US, LSIL, HSIL, or Unsatisfactory).
  Outcome Measurement Tool: Liquid-based cytology (ThinPrep) interpreted using the 2014 Bethesda System.
  Unit of measure:
  Percentage of participants
Correlation Between Participant Characteristics and Abnormal Cytology | At time of screening
  Correlation between participant demographic & clinical factors (age, parity, contraceptive use, comorbidities) and presence of abnormal cytology.
  Unit of measure:
  Correlation coefficient (r)
  Measurement tool:
  Statistical analysis (Pearson/Spearman correlation)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M El-Minawi, Professor, Principal Investigator — Cairo University; Yossra Lasheen, Assistant Professor, Study Chair — Cairo University; Mohamed Aly, Lecturer, Study Director — Cairo University
Locations (1):
- Kasr Al-Aini Hospital - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The study does not plan to share individual participant data. The collected data contain identifiable clinical information and cervical cytology results, and the ethics approval does not permit public release of raw participant-level data. Aggregated data may be available upon reasonable request.